CLINICAL TRIAL: NCT04461262
Title: A Prospective Multicentre Randomized Study To Assess The Impact Of A Catheter Coating On Clinical Bacteriuria
Brief Title: The Impact Of A Catheter Coating On Clinical Bacteriuria
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Camstent Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Cam-Cath-001
Record Dates: First submitted 2020-07-01; First posted 2020-07-08 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Bacteriuria
MeSH Terms: conditions — Bacteriuria

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Urine samples will not state which arm the participant is in
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Camstent Coated Catheter (Experimental): The patented 'M4D coating' is applied to inner and outer surfaces using a 'dip/dry' process before sterilisation, creating a safe, inert, and long-lasting finish. The coating reduces friction of the catheter surface, enhancing patient comfort on insertion and withdrawal. It also incorporates the materials which virtually preclude biofilm formation. The coating doesn't elute antibacterial agents or toxins, avoiding the build-up of dead bacteria on the device surface and retaining effectiveness throughout extended use (NB. Effectiveness is not lost because of leaching away of an active antimicrobial agent). Finally, the absence of anti-bacterial moieties means that the healthy microbial flora is not disturbed. The device is CE marked
  Interventions: Device: Camstent Coated Catheter
- Standard Care (Other): Foley catheter, uncoated
  Interventions: Device: Standard Care

INTERVENTIONS:
Device: Camstent Coated Catheter — The patented 'M4D coating' is applied to inner and outer surfaces using a 'dip/dry' process before sterilisation, creating a safe, inert, and long-lasting finish. The coating reduces friction of the catheter surface, enhancing patient comfort on insertion and withdrawal. It also incorporates the materials which virtually preclude biofilm formation. The coating doesn't elute antibacterial agents or toxins, avoiding the build-up of dead bacteria on the device surface and retaining effectiveness throughout extended use (NB. Effectiveness is not lost because of leaching away of an active antimicrobial agent). Finally, the absence of anti-bacterial moieties means that the healthy microbial flora is not disturbed. The device is CE marked
  Other Names: Standard Care
  Arms: Camstent Coated Catheter
Device: Standard Care — Uncoated Foley catheter
  Arms: Standard Care

SUMMARY:
A prospective multicentre randomized study to assess the impact of a catheter coating on clinical bacteriuria when compared to an uncoated foley catheter.

Each participant will take part in the trial from the time the participant signs the informed consent form (ICF).

After the screening visit, the participants will be randomized to either a coated catheter or an uncoated catheter. Participants will be assigned to receive trial treatment until the catheter has been removed as per standard hospital guidelines, investigator's decision to withdraw the subject, noncompliance with trial treatment or procedures, unacceptable adverse event, or participant withdraws consent.

During the trial urine samples will be taken form the catheter port, temperature will be taken, and participants and healthcare providers will be asked to complete questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Require insertion or exchange of a catheter as a component of their routine clinical care as per hospital guidelines
2. Patients aged 18+ years will be eligible for the study.
3. Patient understands and is willing to participate in the study and is able to comply with study procedures and visits.

Exclusion Criteria:

1. Patients that have or recently (within 3 weeks) had a urinary catheter and displays symptoms of current urinary tract infection.
2. Pregnant or Breastfeeding.
3. Patients with a potentially immunocompromised conditions (HIV)
4. Has a known silicone allergy or sensitivity
5. Use of investigational drug or device within four weeks prior to study entry that may interfere with this study.
6. Any medication deemed by the Investigator to potentially interfere with the study treatment
7. Participation in any other clinical study.
8. Has a known bloodstream infection or an infection that requires prolonged antibiotic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2021-04-27 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Change in the number of days in which bacterial concentrations are greater than 10^5 CFU/mL in coated catheters, as compared to uncoated control catheters | 1 Year

SECONDARY OUTCOMES:
Change in the number of cases experiencing Symptomatic Bacteriuria (CAUTI) coated catheters vs. uncoated controls | 1 Year
Change in the number of cases receiving prophylactic or therapeutic Antibiotics during catheter use in coated catheters vs. uncoated controls | 1 Year
Patient Reported Outcomes (PRO) | 1 Year
  EQ-5D-5L questionnaire will be given to participants as well as a questionnaire asking participants on their experience using the catheter

CONTACTS AND LOCATIONS:
Overall Officials: Prital Patel, Study Director — Camstent Ltd.
Locations (4):
- United Kingdom (4):
  - Stoke Mandeville Hospital, Buckingham
  - Addenbrookes Hospital, Cambridge
  - Royal National Orthopaedic Hospital, London
  - Norfolk & Norwich University Hospital, Norwich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Camstent — http://camstent.com/